CLINICAL TRIAL: NCT05262712
Title: SFB TRR 169/A3 (2.FP) Crossmodal Learning in Health and Neurological Disease: Neurocomputational Representation and Therapeutic Application (Task 2-2)
Brief Title: Crossmodal Learning in Therapeutic Processes (Task 2-2)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unability to reach anticipated participant numbers during COVID pandemic
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Research Foundation (Other); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFB TRR 169/A3 (2-2)
Record Dates: First submitted 2022-02-05; First posted 2022-03-02 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Sensory Ataxia
Keywords: Vibro-tactile Stimulation; Neurorehabilitation; Ataxia
MeSH Terms: conditions — Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Assessment, motor training, data analyzes and group allocation are done by different persons. Participants as well as the assessor, the trainer and the investigator are blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation (Experimental): During motor training participants in the stimulation arm receive vitro-tactile feedback applied to the feet when touching an object as measured by force-sensing resistors mounted to the sole of the feet.
  Interventions: Device: Vibro-tactile stimulation
- Control (Placebo Comparator): The control group receives the same motor training with the same derives (force-sensing resistors, vibro-tactile stimulators) mounted to the feet but receives no stimulation.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Device: Vibro-tactile stimulation — Vibro-tactile stimulation will be administered to the feet of participants via C2 tactors (diameter: 3.05 cm, height: 0.79 cm, operating frequency: 200-300 Hz see https://www.eaiinfo.com/tactor-info/). Vibro-tactile stimulation will be triggered by force-sensing resistors (TEA CAPTIV T-SENS FSR, see https://www.teaergo.com/products/tea-captiv-t-sens-fsr/).
  Arms: Stimulation
Other: Placebo Control — Devices mounted, no stimulation
  Arms: Control

SUMMARY:
Interventional study of the effects of vibro-tactile feedback on behavioral deficits and learning during motor training in patients with sensory ataxia.

ELIGIBILITY:
Inclusion Criteria:

* Electrophysiological diagnosis of sensory ataxia
* Age >= 18, <=80
* Existing declaration of consent

Exclusion Criteria:

* Pregnancy
* Lacking capacity for consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Timed Up-and Go Test | One day before (baseline) and one day after seven days of motor training
  The Timed "Up and Go" test is a clinical test to assess a patient's mobility and risk of falling.

SECONDARY OUTCOMES:
Change from baseline in 10-Meter-Walk Test | One day before (baseline) and one day after seven days of motor training
  The 10-Meter-Walk Test is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility and gait.
Change from baseline in Berg-Balance-Scale | One day before (baseline) and one day after seven days of motor training
  The Berg-Balance-Scale (BBS) is used to determine a patient's ability to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
Change from baseline in Postural-Sway Test | One day before (baseline) and one day after seven days of motor training
  The Postural-Sway Test is a common test of quiet stance balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Neurologie, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is planned after main publication of results.
Supporting Information: Study Protocol
Time Frame: Within 24 months after main publication.
Access Criteria: Personal login into UKE data repository.